CLINICAL TRIAL: NCT06007742
Title: Parent-administered Pediatric Tuina for Improving Sleep Quality and Appetite in School-aged Children With ADHD: a Pilot Randomized Controlled Trial
Brief Title: Parent-administered Pediatric Tuina for Improving Sleep Quality and Appetite in School-aged Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT_ADHD_AS
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group: parent-administered pediatric tuina (n=20) (Experimental)
  Interventions: Other: parent-administered pediatric tuina
- Active control group: parent-child interactive exercise (n=20) (Active Comparator)
  Interventions: Other: parent-administered pediatric tuina
- Control group: usual care (n=20) (No Intervention)

INTERVENTIONS:
Other: parent-administered pediatric tuina — Parents in intervention group will participate in a pediatric tuina course to improve eating and sleep symptoms of ADHD, followed by an 8-week treatment period for the children. The course will take place at the Hong Kong Polytechnic University campus and will consist of 2 sessions of approximately 2 hours each. The course content will be taught by a registered TCM practitioner.
  . Parents assigned to this group will participate in a Parent-Child Exercise for ADHD program, which will complete with their children in the next 8 weeks. The program will take place at the Hong Kong Polytechnic University campus and will consist of 2 sessions of approximately 2 hours each. The content will be taught by a registered physiotherapist.
  The two intervention groups are manipulated every other day for 25-30 minutes each. A total number of interventions equal to or greater than 24 is considered a completed intervention.
  Other Names: parent-child interactive exercise
  Arms: Active control group: parent-child interactive exercise (n=20); Intervention group: parent-administered pediatric tuina (n=20)

SUMMARY:
Title: Parent-administered pediatric tuina for improving sleep quality and appetite in school-aged children with ADHD: a pilot randomized controlled trial

Background: Pediatric tuina has been used and explored by many researchers and clinicians as a topical complementary and alternative treatment for ADHD, which can compensate for some of the shortcomings of medications and behavioural therapies, such as the side effects of medications and the financial stress of long-term behavioural therapies. Pediatric tuina can also grasp the golden stage of young children and improve their symptoms in time on the basis of TCM pattern identification and holistic concepts. We once conducted a focus group interview on 15 parents to understand the effects of parent-administered pediatric tuina on ADHD symptoms, and all parents reported that parent-administered pediatric tuina significantly improved the child's sleep quality, eating habits, and parent-child relationship within a short period of time after receiving the intervention.

Objective: This study aims to assess the preliminary effects, feasibility, and safety of parent-administered pediatric tuina for attention deficit hyperactivity disorder (ADHD) symptoms in school-aged children.

Methods: This project is a three-arm, parallel, open-label, pilot RCT. Sixty participants were randomized into three groups at a 1:1:1 ratio. Parents in the parent-administered tuina group (n = 20) will attend a face-to-face training program on pediatric tuina for ADHD and conduct this intervention on their children at home. Parents in the parent-child interaction group (n = 20) will attend face-to-face training about parent-child interactive exercises and carry them out with their children at home. Both interventions will be carried out every other day during a two-month intervention period, with each manipulation for at least 25-30 min. Participants in the waitlist group (n=20) will not receive both interventions during the intervention period. Outcomes will be assessed at baseline, week 4, and week 8. The primary outcome measure was the Sleep Disturbance Scale for Children; the secondary outcomes included Children's Eating Behaviour Questionnaire, Conners Parent Rating Scale, and Child Health Questionnaire. A process evaluation will be embedded within the outcome evaluation. Descriptive statistics for sociodemographic variables and clinical variables will be presented. Data will be presented as mean and standard deviation. The feasibility outcomes will be presented as percentages. The rating scale scores between the intervention groups and the control group in week 4 and week 8 will be compared using a linear mixed-effects model. Recorded interviews will be transcribed verbatim and analyzed using content analysis. Depending on the topic and purpose of the study, the interview was categorized into words or sentences with the help of the qualitative research tool Nvivo.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the children are the following:

  1. Children: Aged 6-8 years old by the start of the assessment (according to the Hong Kong Education Bureau, 6 years old is considered suitable for primary school education)
  2. Have an internationally recognized diagnosis or documentation of ADHD
  3. Have a score of more than 39 on the Sleep Disturbance Scale for Children (SDSC)
* Inclusion criteria for the parents are the following

  1. Ability to communicate in Cantonese
  2. Willingness to learn the knowledge and manipulations of pediatric tuina for ADHD symptoms
  3. Available to visit the Hong Kong Polytechnic University to attend the course as scheduled in accordance with the trial process
  4. Sign the informed consent form

Exclusion Criteria:

* Exclusion criteria for the children are the following:

  1. Currently receiving other tuina (or massage) treatments
  2. Having other developmental disorders (e.g., autism, intellectual disability)
  3. Having acute infectious diseases (e.g., scarlet fever, chicken pox, etc.), hemorrhagic diseases (e.g., bleeding, local places of various kinds of malignant tumor), or dermatological problems (e.g., scald, severe skin lesion, skin infections)
  4. Having any severe illness or medical condition (e.g., fractures, paraplegia) that are not suitable to receive pediatric tuina
* Exclusion criteria for the parents are the following:

  1. Having any severe psychiatric disorder (e.g., major depression)
  2. Having difficulties to conduct massage therapy due to physical problems
  3. Having a score less than 22 on the Montreal Cognitive Assessment (MoCA).

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Disturbance Scale for Children (SDSC) Chinese version | Baseline, week 4, and week 8.
  The SDSC is a 26-item scale used to evaluate specific sleep disturbance in children. The scale is divided into 6 dimensions, representing 6 types of sleep disturbance: disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhydrosis. Each item is scored on a 5-point Likert scale from 1-5. The higher the total score, the more serious the sleep disturbance is, and a total score of more than 39 is considered to be a sleep disturbance.

SECONDARY OUTCOMES:
Children's Eating Behaviour Questionnaire (CEBQ) Chinese version | Baseline, week 4, and week 8.
  The Child Eating Behavior Questionnaire (CEBQ) is a 35-item parent-report questionnaire assessing eating style in children. Eating style is assessed on eight scales: food responsiveness (4 items), enjoyment of food (4 items), emotional overeating (4 items), desire to drink (3 items), satiety responsiveness (5 items), slowness in eating (4 items), and emotional undereating (4 items), and fussiness (7 items). Informants rate the frequency of their child's behaviors and experiences on a 5-point scale: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always.
Conners Parent Rating Scale (CPRS) Chinese version | Baseline, week 4, and week 8.
  The CPRS is used to assess ADHD in children aged 3-17 years. It assesses the child's behaviour problems, attention deficit disorder, and hyperactivity through the parent's perspective. The scale identifies behavioural problems, learning problems, psychosomatic problems, impulsivity-hyperactivity, and anxiety problems. Each item is rated on a four-point scale: 0-3. The higher the average score, the more significant the problem, and above 1.5, the more likely ADHD is present.
Child Health Questionnaire (CHQ) Chinese version | Baseline, week 4, and week 8.
  The parent-reported CHQ is used to assess the healthy quality of life in children and adolescents aged 5 to 18 years, measuring 14 unique physical and psychological concepts. A 28-item version is used for this study, divided into two subscales: physical and psychosocial, which included 14 basic dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong, China